CLINICAL TRIAL: NCT06636214
Title: Adapting the CHATO Communication Intervention for Diverse Nursing Home Communities
Brief Title: Adapting Changing Talk: Online (CHATO) to CHATO-Inclusive
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Oklahoma (Other); University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01AG085177 (NIH)
Record Dates: First submitted 2024-09-23; First posted 2024-10-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Dementia
Keywords: ADRD; Nursing Home Staff Communication; Elderspeak
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHATO Inclusive Intervention (Experimental)
  Interventions: Behavioral: CHATO-I
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: CHATO-I — Online communication education program
  Arms: CHATO Inclusive Intervention

SUMMARY:
The study will adapt and test the current CHATO training to be more culturally acceptable for nursing homes with diverse staff and residents.

DETAILED DESCRIPTION:
A person is diagnosed with Alzheimer's disease or related dementia (AD/ADRD) every 65 seconds, and most persons living with dementia (PLWD) experience nursing home (NH) care at some stage.Dementia is most prevalent among Black and Hispanic Americans who are increasingly cared for in NHs. NH staff shortages and lack of dementia care skills limit care quality, especially in NHs serving high proportions of minority residents. Care is complicated by the behavioral and psychological symptoms of dementia (BPSD) of PLWD who cannot express their unmet physical and psychosocial needs. BPSD increase staff stress and time to complete care and contribute to staff turnover, injury, and inappropriate psychotropic medication use.

The PI and other researchers have empirically verified that BPSD occur when staff use elderspeak (speech like baby talk) that features inappropriately intimate terms of endearment (diminutives such as "honey"), belittling pronoun substitutions that imply dependence ("we" need a bath), and harsh task-oriented commands ("sit down"). Elderspeak conveys a message of disrespect and incompetence to PLWD who react with withdrawal or BPSD. The investigators R03 study first established that elderspeak use more than doubled the occurrences of resident responses of BPSD (measured by timed sequential behavioral analyses of BPSD in relation to type of staff communication in video data). The investigators R01 trial (NR011455) confirmed that the three-session Changing Talk(CHAT) staff education intervention reduced staff elderspeak use that significantly reduced resident BPSD.The evidence-based CHAT intervention was transitioned to online modules (CHATO), maintaining content, active engagement, and application activities, with equal knowledge gain (mechanism of action) and improved participation and completion rates. The investigators are currently testing CHATO in a pragmatic national trial in 128 NHs (R01AG069171). However, NHs serving high minority-resident populations with fewer resources and staff and more frequent and serious care deficiencies, including high antipsychotic medication use rates, have been less likely to respond to recruitment and study participation. Research has established that tailoring interventions and intensification of recruitment and implementation approaches are frequently necessary to reach and achieve intervention success to overcome health care disparities in diverse care settings.

This study will engage staff from NHs serving diverse residents with an expert stakeholder advisory panel to adapt the content and format of CHATO to the new CHATO-Inclusive (CHATO-I) to increase cultural competency and inclusiveness for diverse NH communities. The investigators will then conduct a cluster randomized trial in NHs (N=40) with high proportions (>25%) of minority residents. NHs will be randomized to intervention or waitlist control groups and one of two waves for staff completion of the tailored CHATO-I intervention with high intensity implementation support. The investigators will test feasibility and acceptability and use hierarchical mixed model analyses to evaluate preliminary effects of the intervention on BPSD and psychoactive medication use in a pragmatic evaluation of NH Electronic Medical Record (EMR) data.

Aim 1 (years 1 and 2): Tailor recruitment, implementation support, and intervention content and format for NHs serving diverse residents. Administrators, directors of nursing, and care staff from six NHs (N=24) serving diverse residents will complete current CHATO and participate in focus groups. Thematic analyses of transcribed recordings will identify tailoring modifications for diverse NH communities. The ADAPT framework will guide adaptation of CHATO to CHATO-I with support from diversity consultants and stakeholders.

Aim 2 (years 3 to 5): Test feasibility, acceptability, and preliminary effects of CHATO-I in 40 NHs serving diverse residents in a cluster-randomized waitlist-controlled trial. Enrollment and completion rates will be used to evaluate feasibility and acceptability (Aim 2a). Mixed modeling will evaluate change in resident BPSD and psychoactive medication use from eight quarters of Minimum Data Set (MDS) and Nursing Home Quality Measure (NHQM) data (Aim 2b). We hypothesize that resident BPSD and psychoactive medication use will be reduced post-CHATO-I.

Aim 3 (years 3 to 5): Validate the mechanism of action of CHATO-I. Additional modeling analyses will evaluate the effects of CHATO-I on learning outcomes (gains in knowledge, confidence, recognition) and intention to use learned skills on resident BPSD and psychoactive medication use. We hypothesize that greater staff knowledge gain and intention to use new skills will be associated with greater outcome reductions.

This Stage 1B research will use the NIA Health Disparities Framework to adapt and expand testing of the evidence-based CHATO intervention for NHs serving diverse resident populations, increasing communication knowledge to reduce health disparities (BPSD and psychotropic medication use). This research addresses the National Plan to Address Alzheimer's disease goals, NIA's milestones for nonpharmacological interventions, and the National Academy National Imperative to improve NH quality through culturally tailored intervention.

ELIGIBILITY:
Inclusion Criteria:

* Medicare certified NHs (N=40) caring for 75% White, non-Hispanic residents, and care for residents diagnosed with AD/ADRD.
* CNAs, nurses, and other direct care staff who are permanent employees of participating NHs and who provide direct care at least 8 hours weekly will complete the CHATO-I training, available by URL link.
* All staff will be encouraged to participate as high staff participation is desired to achieve facility-wide communication change. NHs will provide the number of eligible staff participants.
* Data for residents in participating NHs with AD/ADRD documented on the MDS Active Diagnoses list will be included in the analyses as well as MDS data for: age, sex, race and ethnicity, frailty (MDS-CHESS scale), and level of cognitive function (MDS Cognitive Performance Scale).

Exclusion Criteria:

* NHs serving 25% of residents admitted prior to age 65 will be excluded (screening out NHs serving primarily younger persons with serious mental illnesses).
* CNAs, nurses, and other direct care staff who do not meet the inclusion criteria. Resident Sample.
* Resident data excluded from MDS includes active psychiatric diagnoses (bipolar disorder, major depressive episode, schizophrenia or schizoaffective disorder, mood disorder with psychotic features, psychotic symptoms, hallucinations, or delusions); terminal illness (on hospice); and lack of response to staff (MDS section B).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-08-31 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Test CHATO's effects on Behavioral and Psychological Symptoms of Dementia (BPSD) - Change in MDS E0200 pre/post intervention | pre (3 months) / post (3 months) post intervention
  CMS MDS Quarterly data - E0200 Presence and Frequency of Behavioral Symptoms in the last 7 days; The steps for assessment are to review the medical record, observe the resident in a variety of situations, and interview staff, across all shifts and disciplines. Coding Instruction: Code 0, behavior not exhibited, Code 1, behavior of this type occurred 1-3 days, Code 2, behavior of this type occurred 4-6 days, but less than daily, or Code 3, behavior of this type occurred daily.
Test CHATO's effects on Behavioral and Psychological Symptoms of Dementia (BPSD) - Change in MDS E0800 pre/post intervention | pre (3 months) / post (3 months) post intervention
  CMS MDS Quarterly data - E0800 Rejection of Care - Presence and Frequency over past 7 days; The steps for assessment are to review the medical record, observe the resident in a variety of situations, and interview staff, across all shifts and disciplines. If the resident exhibits behavior that appears to communicate a rejection of care (and that rejection behavior has not been previously determined to be consistent with the resident's values or goals), ask him or her directly whether the behavior is meant to decline or refuse care. Coding Instruction: Code 0, behavior not exhibited, Code 1, behavior of this type occurred 1-3 days, Code 2, behavior of this type occurred 4-6 days, but less than daily, or Code 3, behavior of this type occurred daily.
Test CHATO's effects on Behavioral and Psychological Symptoms of Dementia (BPSD) - Change in MDS E1100 pre/post intervention | pre (3 months) / post (3 months) post intervention
  CMS MDS Quarterly data - E1100 Change in Behavioral or Other Symptoms: The steps for assessment are review responses provided to items E0100-E1000 on the current MDS assessment, compare with responses provided on prior MDS assessment, and then taking all of these MDS items into consideration, make a global assessment of the change in behavior from the most recent to the current MDS. Rate the overall behavior as same, improved, or worse.
  Coding Instructions: Code 0, same: if overall behavior is the same (unchanged), Code 1, improved: if overall behavior is improved, Code 2, worse: if overall behavior is worse, or Code 3, N/A: if there was no prior MDS assessment of this resident.
Test CHATO's effects on psychotropic medication - Change in MDS N0410 pre/post intervention | pre (3 months) / post (3 months) post intervention
  CMS MDS Quarterly data - N0410 Medications Received: The steps for assessment are review the resident's medical record for documentation that any of these medications were received by the resident during the 7-day look-back period (or since admission/entry or reentry if less than 7 days) and review documentation from other health care settings where the resident may have received any of these medications while a resident of the nursing home (e.g., valium given in the emergency room). Coding Instructions: N0410A, Antipsychotic,N0410B, Antianxiety, N0410C, Antidepressant, N0410D, Hypnotic, N0410E, Anticoagulant, N0410F, Antibiotic, N0410G, Diuretic
Test CHATO's effects on psychotropic medication - Change in NHQM Prescribed Antipsychotic pre/post intervention | pre (3 months) / post (3 months) post intervention
  CMS Quarterly Nursing Home Quality Measure: Prescribed Antipsychotic (Long-stay quality measure 419) The percentage of long-stay residents who are receiving antipsychotic drugs in a 7-day look-back period. Exclusions: Residents with a diagnosis of schizophrenia, Tourette's syndrome, or Huntington's disease. Reported by nursing homes quarterly and gathered from Nursing Home Compare.
Test CHATO's effects on psychotropic medication - Change in Survey 757 and 758 Noncompliance | pre (3 months) / post (3 months) post intervention
  Survey 757 and 758 (prior 319), Noncompliance due to unnecessary medications and level of deficiency - Noncompliance due to unnecessary medications and level of deficiency (immediate jeopardy, actual harm, no actual harm & isolated, pattern and occurrence).

SECONDARY OUTCOMES:
Analyze NH strategies to engage staff and maximize CHATO effects _ Change in Knowledge at post intervention | post intervention
  CHAT Scale - 13 questions, measures knowledge gained from training. Scale would be 0-13, Higher scores indicate more knowledge gained and better outcomes. During Aim 1 of the grant, we will determine a new time frame for the intervention.
Analyze NH strategies to engage staff and maximize CHATO effects _ Change in Communication Ratings | post intervention
  Communication Rating Sheet - Participant watches a video and answers questions testing their ability to visually and audibly identify effective vs ineffective communication strategies and recognize elderspeak vs. person-centered care. During Aim 1 of the grant, we will determine a new time frame for the intervention.
Analyze NH strategies to engage staff and maximize CHATO effects _ Implementation Strategies utilized during the training phase | post intervention
  A descriptive implementation survey created by the investigators will identify the approach types (Implementation Teams, Champions, Stakeholders, Location of training, NH Communication Plan, Discussion Types, and Incentives), motivation to participate in research, and NH level evaluation.During Aim 1 of the grant, we will determine a new time frame for the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Williams, RN, PhD, Principal Investigator — University of Kansas